CLINICAL TRIAL: NCT04514159
Title: A Phase 1b Study of ZN-c5 in Combination With Abemaciclib in Patients With Estrogen-Receptor Positive, Human Epidermal Growth Factor Receptor-2 Negative Advanced Breast Cancer
Brief Title: A Study of ZN-c5 and Abemaciclib in Participants With Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zeno Alpha Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZN-c5-003
Record Dates: First submitted 2020-08-11; First posted 2020-08-14 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Breast Cancer
Keywords: Dose escalation; Phase 1 combination; Selective estrogen receptor degrader; Hormone sensitive; Estrogen receptor; Hormone receptor
MeSH Terms: conditions — Breast Neoplasms | interventions — abemaciclib

STUDY DESIGN:
Intervention Model Description: All participants will receive the same treatment but ZN-c5 will be given at different doses in this dose escalation study.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ZN-c5 + abemaciclib combination therapy (Experimental): Participants will take abemaciclib (150mg) orally twice a day and ZN-c5 (dose escalation) orally once or twice a day to determine the safety, tolerability, and maximum tolerated dose (MTD) or recommended Phase 2 dose (RP2D).
  Interventions: Drug: ZN-c5; Drug: Abemaciclib

INTERVENTIONS:
Drug: ZN-c5 — ZN-c5 is the study drug.
Drug: Abemaciclib — Abemaciclib (VERZENIO®) is an approved drug.
  Other Names: VERZENIO®

SUMMARY:
This is a Phase 1b, open-label, multicenter, dose-escalation study to evaluate the safety, tolerability, pharmacokinetics (PK), and preliminary efficacy of ZN-c5 administered orally in combination with abemaciclib (VERZENIO®) in participants with advanced estrogen-receptor positive, human epidermal growth factor receptor-2 negative (ER+/HER2-) breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age
* Women can be peri- or postmenopausal, as defined by at least one of the following:

  * Age ≥ 60 years;
  * Age < 60 years and cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; and serum estradiol and follicle-stimulating hormone (FSH) level within the laboratory's reference range for postmenopausal females;
  * Documented bilateral oophorectomy;
  * Must receive a gonadotrophin-releasing hormone agonist beginning at least 4 weeks prior to the first dose of study medication
* Histologically or cytologically confirmed diagnosis of advanced adenocarcinoma of the breast
* Estrogen receptor positive disease
* Human Epidermal Growth Factor Receptor 2 negative disease
* Measurable disease per Response Evaluation Criteria in Solid Tumors v1.1

Exclusion Criteria:

* Prior therapy within the following windows:

  * Tamoxifen, aromatase inhibitor, fulvestrant, or other anti-cancer endocrine therapy < 14 days;
  * Any investigational drug therapy < 28 days or 5 half-lives (whichever is shorter)
  * Any prior systemic chemotherapy regardless of the stop date, but the subject must have recovered to eligibility levels from prior toxicity
* Prior treatment with CDK4/6 inhibitors
* Unexplained symptomatic endometrial disorders (including, but not limited to, endometrial hyperplasia, dysfunctional uterine bleeding, or cysts)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2022-10-24 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events from ZN-c5 in combination with abemaciclib | Through study completion, anticipated to be 21 months
  Measured by the number of treatment-emergent adverse events and graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0

SECONDARY OUTCOMES:
Determine tumor responses to combination treatment | Through study completion, anticipated to be 21 months
  Measured by radiographic responses as defined by revised Response Evaluation Criteria in Solid Tumor (RECIST) v1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Carrie Brownstein, MD, Study Chair — Zeno Alpha Inc.
Locations (5):
- United States (2):
  - Site 2, Gilbert, Arizona
  - Site 1, Charleston, South Carolina
- Poland (3):
  - Site 6, Grudziądz
  - Site 4, Krakow
  - Site 5, Lodz